CLINICAL TRIAL: NCT04234009
Title: The Effects of a Healthy Lifestyle Intervention on Brain Vascular Function in Older People
Brief Title: Lifestyle and Brain Vascular Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not possible due to COVID-19
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: METC19-072
Record Dates: First submitted 2019-12-20; First posted 2020-01-21 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy Lifestyle; Physical Exercise; Healthy Diet; Cerebrovascular Circulation; Cerebral Blood Flow; Glucose Metabolism; Cognitive Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy lifestyle (Experimental): Healthy lifestyle intervention, which includes physical activity and dietary advice according to the dutch guidelines.
  Interventions: Other: Healthy Lifestyle
- Control (No Intervention): Maintenance of habitual physical activity and diet

INTERVENTIONS:
Other: Healthy Lifestyle — The physical activity guidelines for older consist of 150 minutes per week moderate-to-high intensity exercise, two times per week muscle and bone strengthening exercises, which are combined with balance exercises. Additional health benefits can be achieved with a longer exercise duration, frequency and/or intensity. Furthermore, the amount of time sitting should be minimised. The dietary guidelines are described in detail in the so-called "The Wheel of Five". In brief, the circle is divided into four food groups and one beverage group. More than half of the circle is covered by fruits, vegetables, whole grain (containing) breads, cereals and potatoes. A much smaller part is compromised by animal source foods, spreads and cooking fats. Water, tea and coffee without sugar complete the circle.
  Arms: Healthy lifestyle

SUMMARY:
Cognitive performance is negatively related to an impaired glucose metabolism, possibly due to impairments in brain vascular function. Supported by the statement from the American Heart and Stroke Association that a healthy lifestyle is one of the most effective strategies to protect against cognitive decline, the investigators now hypothesise that healthy lifestyle intervention-induced changes in glucose metabolism cause beneficial effects on brain vascular function thereby improving cognitive performance. The primary objective of this intervention study is thus to evaluate in sedentary older men and women the effect of a 16-week aerobic-based exercise program on cerebral blood flow, as quantified by the non-invasive gold standard magnetic resonance imaging (MRI) perfusion method Arterial Spin Labeling (ASL). Cerebral blood flow is a robust and sensitive physiological marker of brain vascular function. Secondary objectives are to examine effects on glucose metabolism using the homeostatic model assessment for insulin resistance (HOMA-ir) and cognitive performance as assessed with a neurophysiological test battery.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-35 kg/m2
* Sedentary (assessed as low physically active using the International Physical Activity Questionnaire)
* Right handedness and footedness
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* Consumption of more than 21 alcoholic units/week (men), or more than 14 alcoholic units/week (women)
* Use of dietary supplements known to interfere with the main study outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging, including permanent facial makeup, surgical clips/material in body, metal splinter in eye or claustrophobia

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Brain vascular function | Baseline (0 weeks)
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)
Brain vascular function | After intervention (16 weeks)
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)

SECONDARY OUTCOMES:
Cognitive performance | Baseline (0 weeks) and after intervention (16 weeks)
  Cambridge Neuropsychological Test Automated Battery (CANTAB)
Glucose metabolism | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Homeostatic Model Assessment for Insulin Resistance (HOMA-ir) and HbA1c

OTHER OUTCOMES:
Flow-Mediated Vasodilation (FMD) | Baseline (0 weeks) and after intervention (16 weeks)
  Peripheral vascular function, endothelial function
Carotid Artery Reactivity (CAR) | Baseline (0 weeks) and after intervention (16 weeks)
  Peripheral vascular function, endothelial function
Pulse Wave Analysis (PWA) | Baseline (0 weeks) and after intervention (16 weeks)
  Peripheral vascular function, vascular stiffness
Pulse Wave Velocity (PWV) | Baseline (0 weeks) and after intervention (16 weeks)
  Peripheral vascular function, vascular stiffness
Retinal microvascular calibers | Baseline (0 weeks) and after intervention (16 weeks)
  Peripheral vascular function, microcirculation
Blood pressure (systolic, diastolic and mean pressure) | Baseline (0 weeks) and after intervention (16 weeks)
  Office and 24-hour ambulatory blood pressure
Serum lipid profile concentration | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Concentration of serum lipids
Serum insulin concentration | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Concentration of insulin in serum
Plasma glucose concentration | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Concentration of glucose in plasma
Homeostatic Model Assessment for Insulin Resistance (HOMA-ir) | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  HOMA-ir is a method used to quantify insulin resistance and beta-cell function
Circulating markers for low-grade systemic inflammation | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Markers for low-grade systemic inflammation (IL-6, TNF-alpha)
Circulating markers for microvascular function | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Markers for microvascular function (sCAM-1, vWf, cGMP)
Circulating marker of neurogenesis | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Brain-derived neurotrophic factor (BDNF)
Glycated haemoglobin (HbA1C) | Baseline (0 weeks) and after intervention (16 weeks)
  HbA1C is a form of hemoglobin (abbreviated Hb) that is chemically linked to a sugar.
Aerobic fitness | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Incremental exhaustive exercise test (Maximal oxygen consumption and power output)
Physical fitness (1) | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Incremental exhaustive exercise test (Maximal Power output)
Physical fitness (2) | Baseline (0 weeks) and after intervention (16 weeks)
  The 6-minute walk test (6 MWT)
Activity monitoring | Baseline (0 weeks) and after intervention (16 weeks) for four consecutive days
  activPAL activity monitor
Self reported physical activity | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  The International Physical Activity Questionnaire
Food frequency questionnaire | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Self reported food consumption
Dutch Healthy Diet index 2015 | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Compliance to the Dutch dietary guidelines based on the FFQ
Quality of Life score | Baseline (0 weeks) and after intervention (16 weeks)
  The Quality of life will be assessed using a 32-item questionnaire
Sleep characteristics | Baseline (0 weeks) and after intervention (16 weeks)
  Sleep characteristics will be assessed using the 10-item Pittsburgh Sleep Quality Index
Fat mass | Baseline (0 weeks) and after intervention (16 weeks)
  Body composition measured with whole body air-displacement by the BodPod
Fat free mass | Baseline (0 weeks) and after intervention (16 weeks)
  Body composition measured with whole body air-displacement by the BodPod
Anthropometrics (1) | Baseline (0 weeks) and after intervention (16 weeks)
  Weight
Anthropometrics (2) | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  BMI
Anthropometrics (3) | Baseline (0 weeks), at the middle (8 weeks) and after intervention (16 weeks)
  Waist and hip circumference (ratio)
Structural brain status (1) | Baseline (0 weeks) and after intervention (16 weeks)
  MRI MPRAGE
Structural brain status (2) | Baseline (0 weeks) and after intervention (16 weeks)
  T2FLAIR
Structural brain status (3) | Baseline (0 weeks) and after intervention (16 weeks)
  R2*

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Joris, Dr, Principal Investigator — Maastricht University; Ronald P. Mensink, Dr, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands